CLINICAL TRIAL: NCT03153618
Title: VALIDATE: Virtual Agent Linked Intelligent Disease Assessment Tool Engine
Acronym: VALIDATE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding and proposal withdrawn
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 39175
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: In a two section clinic, the plan is to invite one section of newly enrolled patients coming to clinic for first visit to participate in interacting with VALIDATE while maintaining the standard of care within the other section for similarly matched patients. Parallel allocation design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VALIDATE subjects (Experimental): Will be invited to interact with VALIDATE to determine if they meet referral indications for cancer predisposition assessment.
  Interventions: Other: VALIDATE system
- Control (No Intervention): Current standard of care will be followed

INTERVENTIONS:
Other: VALIDATE system — Will be invited to interact with VALIDATE to answer questions about Family Cancer history and some personal medical and lifestyle history. Based on responses, VALIDATE will determine if they meet referral indications for cancer predisposition assessment.
  Arms: VALIDATE subjects

SUMMARY:
The collection and analysis of family, medical, lifestyle, and environmental exposure history (a Comprehensive Health History or "CHH") can identify critical risk factors for many chronic and life-threatening conditions, including cancer. Despite its importance, CHH is infrequently documented and analyzed in primary-care medical practice due to numerous hurdles, and currently available tools have proven inadequate to address this critical problem. This study will evaluate the Virtual Agent Linked Intelligent Disease Assessment Tool Engine ("VALIDATE") system as an easy to administer, accurate, cost-effective, and clinically useful tool for collecting and analyzing structured CHH data.

DETAILED DESCRIPTION:
Our study's objective is to evaluate the Virtual Agent Linked Intelligent Disease Assessment Tool Engine ("VALIDATE") system as a means to improve the affordability and ease, while maintaining the validity and feasibility, of collecting, assessing, and acting on Comprehensive Health History data.

Virtual Agents (VAs) are fully autonomous and embodied software agents that use both verbal (e.g. speech) and non-verbal modalities (e.g., gaze, gesturing) to simulate a clinician-patient encounter. These agents have already successfully shown advantages to patients for: entering family history data on their own, facilitating medication adherence, providing behavioral health information, serving as clinical interviewers, promoting breastfeeding, and educating about and motivating exercise and weight loss. The VALIDATE system has been developed to be a fully automated alternative to the currently extremely labor-intensive process of collecting and transcribing CHH data. VALIDATE will be evaluated for its capability to significantly diminish clinician time and cost to collect, review, analyze, and document accurate and complete certain CHH data directly from patients at home using their own personal desktop computers. VALIDATE will also be evaluated for its capability to identify valid clinical action, e.g. referral indications for familial cancer assessment based on American College of Medical Genetics and Genomics (ACMG)/National Society of Genetic Counselors (NSGC) and National Comprehensive Care Network (NCCN) Guidelines.

ELIGIBILITY:
Inclusion Criteria:

All adults above the age of 18

Exclusion Criteria:

Children under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants satisfied with usage of VALIDATE | Up to sixteen weeks
  At the end of the session, participants will be asked if 1. they enjoyed the process d 2. if they prefer this process versus completing a web or paper form and 3. would they recommend the process to others?
Concordance of data collection - identified relatives | Up to sixteen weeks
  Accuracy rates will be calculated by dividing the number of VALIDATE identified relatives by the number identified by a trained Clinician
Concordance of data collection - identified cancers | Up to sixteen weeks
  Accuracy rates will be calculated by dividing the number of VALIDATE identified cancers by the number identified by a trained Clinician
Number of VALIDATE subjects versus Control subjects identified for further cancer predisposition assessment. | Up to sixteen weeks

CONTACTS AND LOCATIONS:
Overall Officials: Baldeep Singh, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No